CLINICAL TRIAL: NCT05626946
Title: Does the Intervention of an Advanced Practice Nurse for Nursing Home Residents Aged 75 and Over in the Grand Nancy Area Make it Possible to Reduce the Use of the Emergency Service for These Residents?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Mahmut GUNDESLI MD (Unknown); Manon DUPRE, internship (Unknown)
Responsible Party: Principal Investigator, BOURDAIRE Victoire, Medical Doctor - Hospital Practitioner, Central Hospital, Nancy, France
Other Study IDs: 2022PI165
Record Dates: First submitted 2022-11-14; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Geriatric Health Services
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nursing Home resident from Grand Nancy area with Advanced Practice Nurse intervention: Patients aged 75 years and over, resident in Nursing Home at the time of inclusion, and received at least once in the emergency room of the Nancy Hospital during the period concerned. Inclusion in the group with IPA intervention for Nursing Home residents of the Grand Nancy area where the Advanced Practice Nurse is authorised to intervene.
  Interventions: Other: Observation
- Nursing Home resident outside Grand Nancy area without Advanced Practice Nurse intervention: Patients aged 75 years and over, resident in Nursing Home at the time of inclusion, and received at least once in the emergency room of the Nancy Hospital during the period concerned. Inclusion in the control group for Nursing Home residents outside the Grand Nancy area without the Advanced Practice Nurse intervention.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
The rate of emergency room visits is high at the extremes of age, with patients aged 75 or over accounting for 12% of emergency room visits, and the time they spend there is significantly longer than that of younger patients.

Nursing Home residents represent 14% of these emergency room visits and only 5% of them on average are not hospitalised and return to their original Nursing Home.

A retrospective study of patients aged 75 and over referred to the emergency department of the Nancy Hospital by the Nursing Homes over a six-month period showed that nearly 30% of patients aged 75 and over referred by their Nursing Home were rehospitalized during the period studied, 1/3 for the same reason and 2/3 for other reasons.

The intervention of an Advanced Practice Nurse (IPA) attached to geriatric practice, among other things, as an interface between Nursing Home and the hospital therefore seems to have its place in improving the care pathway for the elderly.

The assessment by an Advanced geriatric Practice Nurse of residents of Nursing Home aged 75 and over in Grand Nancy area one week after a visit to the emergency room significantly reduces the number of new visits to the emergency room by these residents over a follow-up period of seven months, compared with residents of Nursing homes aged 75 and over (outside Grand Nancy area) who do not benefit from an assessment by an Advanced Practice Nurse.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information on the organization of the research and has not objected to the use of this data
* Elderly men and women 75 years of age and older at the time of the emergency room visit
* Having for main residence one of the nursing homes
* Administratively present in the emergency department

Exclusion Criteria:

* People under 75 years of age
* Residing at home or in a senior residence
* Referred by an inpatient department (rehabilitation department)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All persons aged 75 and over, residents of nursing homes ,who consulted the emergency department of Nancy Hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
RATE OF REHOSPITALISATION OVER THE ENTIRE FOLLOW-UP PERIOD IN THE 2 GROUPS OF PATIENTS WITH AND WITHOUT ADVANCED PRACTICE NURSE INTERVENTION | through study completion, an average of 7 months

SECONDARY OUTCOMES:
PROPORTION OF AVOIDABLE VISITS FOR A REASON SIMILAR TO THE REASON FOR INITIAL HOSPITALISATION | through study completion, an average of 7 months
PROPORTION OF PATIENTS DIRECTLY ADMITTED TO THE NANCY HOSPITAL GERIATRIC UNIT | through study completion, an average of 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France